CLINICAL TRIAL: NCT05662553
Title: A Prospective, Multi-center, Randomized Controlled Clinical Study of ENB Guided MWA Combined With VATS Versus Sequential Surgery for Synchronous Bilateral Multiple Primary Lung Nodules
Brief Title: ENB Guided MWA Combined With VATS Versus Sequential Surgery for Synchronous Bilateral Multiple Primary Lung Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Tang-Du Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-016
Record Dates: First submitted 2022-11-28; First posted 2022-12-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Multiple Primary Lung Cancer
Keywords: electromagnetic navigation bronchoscopy; microwave ablation; sequential surgery
MeSH Terms: interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation (Experimental): After randomization, the enrolled patients in this arm should be performed path simulation under ENB with preoperative CT. On the operation day, single-cavity intubation will be carried out first, and the secondary lesion will be reached through the planned path. After that，the biopsy tissue of the lesion will be sent to ROSE for detection. If malignant，the ablation will be performed，and the location, energy and ablation time will be adjusted according to intraoperative CT. After ablation, radical surgery will be performed on the primary lesion.
  Interventions: Procedure: ENB guided MWA combined with VATS
- Surgery (Active Comparator): The control group will undergo VATS treatment on the primary lesion on the day of operation, and will be re-admitted to the hospital after discharge and recovery (3-4 months) for contralateral secondary lesion surgery.
  Interventions: Procedure: sequential surgery

INTERVENTIONS:
Procedure: ENB guided MWA combined with VATS — ENB guide MWA combine ENB, microwave ablation and 3D reconstruction technology, and guide the probe in the airway to the target lesion for ablation therapy, which is safe and effective. For patients with synchronous bilateral multiple primary pulmonary nodules, ENB guide MWA combined with VATS treatment can not only avoid the risk of bilateral surgery, but also complete the "one-stop" treatment, which is a new treatment mode.
  Arms: Ablation
Procedure: sequential surgery — Bilateral surgery is a traditional treatment, but it will lead to increased intraoperative risk and postoperative complication rate, and more likely to lead to postoperative complications such as decreased quality of life and cardiopulmonary dysfunction.
  Arms: Surgery

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of ENB guided MWA combined with VATS versus sequential surgery for synchronous bilateral multiple primary lung nodules. Participants will be divided into two group.One group will accepte treatment of ENB guided MWA combined with VATS,another will accepted sequential surgery.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancers and the leading cause of cancer-related death worldwide. With the improvement of people's health awareness and the wide application of LDCT and HRCT, the incidence of multiple primary lung cancer is increasing, especially the synchronous bilateral multiple primary pulmonary nodules are the difficulties in the treatment of pulmonary nodules. Bilateral sequential surgery is associated with higher intraoperative risks, higher rates of postoperative complications, and lower postoperative quality of life. At present, a small number of recent retrospective studies have shown that microwave ablation(MWA) guided by electromagnetic navigation bronchoscopy(ENB) combined with video-assisted thoracic surgery(VATS) treatment can effectively treat bilateral multiple primary pulmonary nodules, which not only has a low complication rate, but also can avoid secondary surgery.

Based on previous studies, the research plans to conduct a prospective, multi-center, randomized controlled study to evaluate the safety and efficacy of ENB guided MWA combined with VATS versus sequential surgery for synchronous bilateral multiple primary lung nodules, as well as its potential value as a new treatment option for these participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years and ≤80 years;
2. The subjects are diagnosed synchronous bilateral multiple primary lung nodules by HRCT
3. The primary nodule is diagnosed as lung cancer by preoperative puncture or multidisciplinary discussion, which can be treated with radical surgery.
4. At least one secondary lesion (6mm≤diameter≤20mm, CTR<0.5) is contralateral to the primary nodule，which need treatment after multidisciplinary discussion
5. The ipsilateral secondary lesions can be treated by sublobar resection at the same time
6. ECOG PS score 0-1
7. The subjects participate voluntarily and sign a written informed consent;

Exclusion Criteria:

1. Patients have contraindications of surgery or anesthesia
2. Patients are unable to undergo bronchoscopy
3. A contralateral secondary lesion is unreachable during ENB planning
4. There are large blood vessels 2 mm near the contralateral secondary lesion
5. Patients have severe bleeding tendency and coagulation dysfunction which cannot be improved in a short time
6. Patients have interstitial pneumonia, pulmonary fibrosis, or severe emphysema
7. Patients have diseases,like severe anemia, dehydration, severe nutritional and metabolic disorders, which cannot be cured or improved in a short time
8. Patients have severe systemic infection and fever (>38.5°C)
9. Patients have other malignant tumors
10. Patients have participated in other clinical trials
11. Investigators consider the patient do not fit for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total perioperative complication rates | From the time of treatment to one month after operation
  Complications refer to operation-related adverse events during and after the operation according to the Clavien-Dindo Classification, including pulmonary infection, Broncho-pulmonary hemorrhage, respiratory failure, pleural effusion, pneumothorax, persistent lung leak, arrhythmia, wound infection, death.

SECONDARY OUTCOMES:
Objective response rate(ORR) | One and three months after ablation
  Objective response rate（ORR）is the proportion of patients with complete responses and partial responses.
Treatment-related side effects | From the time of treatment to one month after operation
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0.
The operation time | During operation
  the duration of the operation in minutes.
The intraoperative blood loss | During operation
  the volume of blood loss in ml.
Postoperative hospital stay (days) | One months after treatment
  The time of hospitalization in days.
Postoperative extubation time (days) | One months after treatment
  The duration of chest drainage in days.
Mortality within 30 days after surgery | One month after treatment
  number of death within 30 days after surgery.
Complications (grade ≥3) | One and three months after treatment
  complications above grade 3 that need to be treated during and after the operation according to the Clavien-Dindo Classification.
Life expectancy(EORTC QLQ-LC29) | One and three months and every year after treatment
  patients' quality of life by questionnaires according to EORTC QLQ-LC29.
Lung function | One and three months and every year after treatment
  forced expiratory volume in one second(FEV1).
3-year disease-free survival(DFS) | A follow-up period of 3 years
  DFS : the time from surgical resection to clinically confirmed local recurrence, distant metastasis, second primary tumor diagnosis, or patient death (control group since the second operation).
The proportion of completed two operations | During operation, an average of 4 months
  the patients in control group complete two operations
The overall cost of treatment | During hospitalization, an average of 2 weeks
  The overall cost of treatment include direct and indirect costs. Additional costs for hospitalization and surgery.

OTHER OUTCOMES:
Biopsy success rate | During operation
  The percentage of people with successful biopsy.
Biopsy positive rate | During operation
  The proportion of patients with malignant biopsies in the overall population

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng LI, PhD, MD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No